CLINICAL TRIAL: NCT01451710
Title: The Effectiveness of Enough Steroids as Inducement Therapy in Minimal Change Disease-like IgA Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, M.D., Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1102
Record Dates: First submitted 2011-10-07; First posted 2011-10-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: IgA Nephropathy
Keywords: enough steroids; MCD; efficacy
MeSH Terms: conditions — Glomerulonephritis, IGA; Macular dystrophy, corneal type 1 | interventions — Prednisone; Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prednisone or Prednisolone (Experimental)
  Interventions: Drug: Prednisone or Prednisolone

INTERVENTIONS:
Drug: Prednisone or Prednisolone — daily single dose of 1mg/kg (maximum 80mg) or alternate day single dose of 2mg/kg (maximum 120mg),maintained for a minimum period of 6 weeks and maximum period of 12 weeks. After achieving complete remission., corticosteroids should be tapered slowly, 10mg every two weeks tapered to reach 0.15mg/kg/d, then 2.5mg every two to four weeks tapered to reach the minimum dosage 10mg/ alternate day
  Other Names: Prednisone, prednisolone, corticosteroids

SUMMARY:
This is a single center,prospective,no-controlled clinical trial

DETAILED DESCRIPTION:
1. The complete remission of enough steroids as inducement therapy in adult minimal change disease-like IgA nephropathy patients
2. The safety of enough steroids as inducement therapy in adult minimal change disease-like IgA nephropathy patients

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged between 18 to 65 years
* Renal biopsy was used to diagnose IgA nephropathy
* Patients with 24h proteinuria 3.5g and serum albumin concentration lower than 30g/L

Exclusion Criteria:

* Patients with serum creatinine ≥ 3 mg/dl or eGFR < 30ml/min per 1.73 m2
* urine RBC > 1 million/ml
* Patients who have received treatment of enough steroids for more than 12 weeks
* patients with secondary IgA
* Patients who have impaired liver function,with ALT/GPT or AST/GOT twice more than the normal upper limit or who have active hepatitis
* Patients with 2 type diabetes or obesity, whose BMI is more than 28kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
24h urinary protein excretion | 3 months

SECONDARY OUTCOMES:
remission rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD, Study Director — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wang J, Juan C, Huang Q, Zeng C, Liu Z. Corticosteroid therapy in IgA nephropathy with minimal change-like lesions: a single-centre cohort study. Nephrol Dial Transplant. 2013 Sep;28(9):2339-45. doi: 10.1093/ndt/gft211. Epub 2013 Jun 19. PMID 23787555